CLINICAL TRIAL: NCT03032172
Title: An Open-Label Study to Investigate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of Risdiplam (RO7034067) in Adult and Pediatric Patients With Spinal Muscular Atrophy
Brief Title: A Study of Risdiplam (RO7034067) in Adult and Pediatric Participants With Spinal Muscular Atrophy
Acronym: Jewelfish
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP39054; 2016-004184-39 (EudraCT Number); 2023-506739-14-00 (EU CTIS Number)
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Risdiplam (Experimental): Participants will receive multiple doses of risdiplam orally once daily for 24 months. After 24-month treatment, participants will be offered the opportunity to enter the open-label extension (OLE) phase for 3 years.
  Interventions: Drug: Risdiplam

INTERVENTIONS:
Drug: Risdiplam — Risdiplam will be administered orally once daily.
  Other Names: RO7034067

SUMMARY:
This is a multi-center, exploratory, non-comparative, and open-label study to investigate the safety, tolerability, PK, and PK/PD relationship of risdiplam in adults, children and infants with Spinal Muscular Atrophy (SMA) previously enrolled in Study BP29420 (Moonfish) with the splicing modifier RO6885247 or previously treated with nusinersen, olesoxime or AVXS-101.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of 5q-autosomal recessive SMA
* Previous enrollment in Study BP29420 (Moonfish) with the splicing modifier RO6885247 or previous treatment with any of the following: 1.) Nusinersen (defined as having received >= 4 doses of nusinersen, provided that the last dose was received >= 90 days prior to screening) or 2.) Olesoxime (provided that the last dose was received <= 12 months and >= 90 days prior to screening) or 3.) AVXS-101 (provided that the time of treatment was >= 12 months prior to screening)
* Adequately recovered from any acute illness at the time of screening and considered well enough to participate in the opinion of the Investigator
* For women of childbearing potential: negative blood pregnancy test at screening, agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating eggs for at least 28 days after the final dose of study drug
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm
* For participants aged 2 years or younger at screening: 1.) Parent or caregiver of participant is willing to consider nasogastric, naso-jejunal or gastrostomy tube placement, as recommended by the Investigator, during the study to maintain safe hydration, nutrition and treatment delivery; 2.) Parent or caregiver of participant is willing to consider the use of non-invasive ventilation, as recommended by the Investigator during the study

Exclusion Criteria:

* Inability to meet study requirements
* Concomitant participation in any investigational drug or device study
* Previous participation in any investigational drug or device study within 90 days prior to screening, or 5 half-lives of the drug, whichever is longer with the exception of studies of olesoxime, AVXS-101, or nusinersen
* Any history of gene or cell therapy, with the exception of AVXS-101
* Unstable gastrointestinal, renal, hepatic, endocrine, or cardiovascular system diseases as considered to be clinically significant by the Investigator
* Inadequate venous or capillary blood access for the study procedures, in the opinion of the Investigator
* For patients aged < 2 years, hospitalization for a pulmonary event within 2 months prior to screening and pulmonary function not fully recovered at the time of screening
* Lactating women
* Suspicion of regular consumption of drugs of abuse
* For adults and adolescents only, positive urine test for drugs of abuse or alcohol at screening or Day -1 visit
* Presence of clinically significant electrocardiogram (ECG) abnormalities before study drug administration from average of triplicate measurement or cardiovascular disease
* History of malignancy if not considered cured
* For participants aged > 6 years, significant risk for suicidal behavior, in the opinion of the Investigator as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Any major illness within one month before the screening examination or any febrile illness within one week prior to screening and up to first dose administration
* Recently initiated treatment for spinal muscular atrophy (within <6 weeks prior to enrollment) with oral salbutamol or another beta 2-adrenergic agonist taken orally
* Any prior use of chloroquine, hydroxychloroquine, retigabin, vigabatrin or thioridazine, is not allowed
* Ascertained or presumptive hypersensitivity (e.g., anaphylactic reaction) to risdiplam or to the constituents of its formulation
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study
* Recent history (less than one year) of ophthalmological diseases
* Any prior use of an inhibitor or inducer of FMO1 or FMO3 taken within 2 weeks (or within 5 elimination half-lives, whichever is longer) prior to dosing

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 174 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- United States (4):
  - Stanford University Medical Center, Palo Alto, California
  - Nemours Children's Hospital, Orlando, Florida
  - Boston Childrens Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- France (5):
  - Hopital Femme Mere Enfant, Bron
  - Hopital Roger Salengro, Lille
  - CHRU de Montpellier, Hopital Gui de Chauliac, Montpellier
  - Hôpital Necker-Enfants Malades, Paris
  - Hopital des Enfants, Toulouse
- Germany (2):
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
- Italy (5):
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Policlinico Agostino Gemelli, Rome, Lazio
  - IRCCS Istituto Giannina Gaslini, Genoa, Liguria
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - UOSD Malattie Neurodegenerative, Messina, Sicily
- UMC Utrecht, Utrecht, Netherlands
- Klinika Neurologii I Wydzialu Lekarskiego WUM w Warszawie, Warsaw, Poland
- Universitäts-Kinderspital (UKBB) Neuropädiatrie, Basel, Switzerland
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - UCL Institute of Child Health & Great Ormond Street Hospital for Children, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Cleary Y, Kletzl H, Grimsey P, Heinig K, Ogungbenro K, Silber Baumann HE, Frey N, Aarons L, Galetin A, Gertz M. Estimation of FMO3 Ontogeny by Mechanistic Population Pharmacokinetic Modelling of Risdiplam and Its Impact on Drug-Drug Interactions in Children. Clin Pharmacokinet. 2023 Jun;62(6):891-904. doi: 10.1007/s40262-023-01241-7. Epub 2023 May 6. PMID 37148485
- See also: roche-sma-clinicaltrials.com provides information about the Roche Jewelfish clinical trial NCT03032172 and molecule being investigated in SMA. — http://roche-sma-clinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 174 adult and pediatric participants with spinal muscular atrophy (SMA) took part in the study at 24 investigative sites across 9 countries from 03 March 2017 to 07 February 2025.
Pre-assignment Details: This study included a 2-year treatment period followed by a 3-year open-label extension (OLE) period. Participants previously enrolled in Study BP29420 (NCT02240355) (Moonfish) and treated with the splicing modifier RO6885247 or previously treated with nusinersen, onasemnogene abeparvovec (AVXS-101), or olesoxime, were enrolled to receive risdiplam. 1 participant previously treated with 'Olesoxime' discontinued per physician's decision before receiving any treatment.
Groups:
- Treatment Phase: RO6885247: Participants previously treated with the splicing modifier, RO6885247 or placebo in study BP29420, received risdiplam, orally (PO), once daily (QD), based on their body weight and age during the 24-month treatment phase.
- Treatment Phase: Nusinersen: Participants previously treated with nusinersen, received risdiplam, PO, QD, based on their body weight and age during the 24-month treatment phase.
- Treatment Phase: Olesoxime: Participants previously treated with olesoxime, received risdiplam, PO, QD, based on their body weight and age during the 24-month treatment phase.
- Treatment Phase: AVXS-101: Participants previously treated with AVXS-101, received risdiplam, PO, QD, based on their body weight and age during the 24-month treatment phase.
- OLE Phase: RO6885247; OLE Phase: Nusinersen; OLE Phase: Olesoxime; OLE Phase: AVXS-101: After the 24-month treatment phase, participants who chose to enter the OLE phase continued receiving risdiplam, PO, QD, based on their body weight and age up to a maximum of 3 years.
Period: Treatment Period
Arm/Group | Treatment Phase: RO6885247 | Treatment Phase: Nusinersen | Treatment Phase: Olesoxime | Treatment Phase: AVXS-101 | OLE Phase: RO6885247 | OLE Phase: Nusinersen | OLE Phase: Olesoxime | OLE Phase: AVXS-101
Started | 13 | 76 | 71 | 14 | 0 | 0 | 0 | 0
Safety-evaluable (SE) Population (SE population included all participants who received at least one dose of risdiplam, whether prematurely withdrawn from the study or not. 1 participant previously treated with 'Olesoxime' discontinued per physician's decision before receiving any treatment and was not included in the SE population.) | 13 | 76 | 70 | 14 | 0 | 0 | 0 | 0
Completed | 11 | 66 | 64 | 13 | 0 | 0 | 0 | 0
Not Completed | 2 | 10 | 7 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance With Study Drug | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinued, but Recorded as Completed Open-label Treatment by the Investigator | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Period: Open-label Extension Period
Arm/Group | Treatment Phase: RO6885247 | Treatment Phase: Nusinersen | Treatment Phase: Olesoxime | Treatment Phase: AVXS-101 | OLE Phase: RO6885247 | OLE Phase: Nusinersen | OLE Phase: Olesoxime | OLE Phase: AVXS-101
Started | 0 | 0 | 0 | 0 | 11 | 66 | 64 | 13
Completed | 0 | 0 | 0 | 0 | 10 | 54 | 49 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 12 | 15 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 7 | 11 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants, regardless of whether they received risdiplam or not.
Groups:
- RO6885247: Participants previously treated with the splicing modifier, RO6885247 or placebo in study BP29420, received risdiplam, PO, QD, based on their body weight and age during the 24-month treatment phase. After the 24-month treatment phase, participants who chose to enter the OLE phase continued receiving risdiplam, PO, QD, based on their body weight and age up to a maximum of 3 years.
- Nusinersen: Participants previously treated with nusinersen, received risdiplam, PO, QD, based on their body weight and age during the 24-month treatment phase. After the 24-month treatment phase, participants who chose to enter the OLE phase continued receiving risdiplam, PO, QD, based on their body weight and age up to a maximum of 3 years.
- Olesoxime: Participants previously treated with olesoxime, received risdiplam, PO, QD, based on their body weight and age during the 24-month treatment phase. After the 24-month treatment phase, participants who chose to enter the OLE phase continued receiving risdiplam, PO, QD, based on their body weight and age up to a maximum of 3 years.
- AVXS-101: Participants previously treated with AVXS-101, received risdiplam, PO, QD, based on their body weight and age during the 24-month treatment phase. After the 24-month treatment phase, participants who chose to enter the OLE phase continued receiving risdiplam, PO, QD, based on their body weight and age up to a maximum of 3 years.
- Total: Total of all reporting groups
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101 | Total
Number analyzed (Participants) | 13 | 76 | 71 | 14 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (14.2) | 16.1 (13.5) | 18.5 (5.7) | 2.5 (1.2) | 17.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 36 | 36 | 3 | 79
  Male | 9 | 40 | 35 | 11 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 6 | 3 | 3 | 12
  Not Hispanic or Latino | 13 | 66 | 63 | 11 | 153
  Unknown or Not Reported | 0 | 4 | 5 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 3 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 11 | 66 | 56 | 10 | 143
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 8 | 12 | 0 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline up to 5 years
Population: SE population included all participants who received at least one dose of risdiplam, whether prematurely withdrawn from the study or not.
Measure: Count of Participants; unit: Participants
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101
Number analyzed (Participants) | 13 | 76 | 70 | 14
Participants | 12 | 76 | 70 | 14

2. Primary Outcome: Number of Participants Who Discontinued Treatment Due to AEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Participants who discontinued treatment due to AEs are reported here.
Time Frame: Baseline up to 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101
Number analyzed (Participants) | 13 | 76 | 70 | 14
Participants | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Shift in Puberty Status From Baseline
Description: Tanner staging of sexual development is a scale used to assess physical maturation as children transition through adolescence into adulthood. Scale defines physical development based on the following characteristics: pubic hair, penis, and testes development in boys; and pubic hair and breast development in girls. It consists of 5 stages, Stage I (prepubertal) to Stage V (mature adult). Participants under 9 years at screening began Tanner staging assessments at 1st visit following their 9th birthday. Tanner data are presented in three categories: Normal (expected stage of puberty based on participant's age at post-baseline visit), Delayed (pubertal development is behind expectations for age at post-baseline visit), & Missing (participant did not attend scheduled visit). Tanner staging assessments were scheduled for participants aged 9-17 years but were also conducted in some older participants, up to age 22. Shift in puberty status from baseline to each week has been represented here.
Time Frame: Baseline, Week 52, 104, 156, 208 and 260
Population: SE population included all participants who received at least one dose of risdiplam, whether prematurely withdrawn from the study or not. Overall number analyzed is the number of participants with data available for analysis. No participants from the AVXS-101 arm were assessed for Tanner staging since all participants in this arm were under 9 years of age.
Measure: Count of Participants; unit: Participants
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101
Number analyzed (Participants) | 4 | 10 | 31 | 0
Participants
  Baseline Status Normal: Week 52 Status Normal | 0 | 0 | 3 |
  Baseline Status Normal: Week 52 Status Missing | 4 | 9 | 27 |
  Baseline Status Delayed: Week 52 Status Normal | 0 | 0 | 1 |
  Baseline Status Missing: Week 52 Status Missing | 0 | 1 | 0 |
  Baseline Status Normal: Week 104 Status Normal | 0 | 4 | 15 |
  Baseline Status Normal: Week 104 Status Missing | 4 | 5 | 15 |
  Baseline Status Delayed: Week 104 Status Missing | 0 | 0 | 1 |
  Baseline Status Missing: Week 104 Status Missing | 0 | 1 | 0 |
  Baseline Status Normal: Week 156 Status Normal | 0 | 0 | 4 |
  Baseline Status Normal: Week 156 Status Missing | 4 | 9 | 26 |
  Baseline Status Delayed: Week 156 Status Missing | 0 | 0 | 1 |
  Baseline Status Missing: Week 156 Status Missing | 0 | 1 | 0 |
  Baseline Status Normal: Week 208 Status Normal | 0 | 0 | 1 |
  Baseline Status Normal: Week 208 Status Missing | 4 | 9 | 29 |
  Baseline Status Delayed: Week 208 Status Missing | 0 | 0 | 1 |
  Baseline Status Missing: Week Status 208 Missing | 0 | 1 | 0 |
  Baseline Status Normal: Week 260 Status Missing | 4 | 9 | 30 |
  Baseline Status Delayed: Week 260 Status Missing | 0 | 0 | 1 |
  Baseline Status Missing: Week 260 Status Missing | 0 | 1 | 0 |

4. Primary Outcome: Number of Participants With Protocol-defined Neurological Conditions (NC)
Description: Neurological examination was performed by asking questions to the participants and/or their caregiver, as well as observing the participants' behavior in general and while performing certain tasks. Questions and tasks were adapted to the age and motor ability of the participant. For very young participants, observing reaction to a sound, speech development, shifting attention to a newly introduced toy, observing the participant interact with the parent/caregiver & for older participants examination of social interaction (school, friends, activities, job as appropriate), memory (e.g., with short word recall), reasoning & language, drawing, etc. Participants with neurological conditions besides those expected with SMA and those expected with SMA are reported.
Time Frame: Baseline up to Week 260
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101
Number analyzed (Participants) | 13 | 76 | 70 | 14
Participants
  Baseline: NC Besides Those Expected With SMA | 0 | 1 | 0 | 1
  Baseline: NC Expected With SMA | 13 | 75 | 70 | 13
  Week 2: NC Besides Those Expected With SMA | 0 | 0 | 0 | 0
  Week 2: NC Expected With SMA | 0 | 3 | 0 | 1
  Week 4: NC Besides Those Expected With SMA | 0 | 0 | 0 | 1
  Week 4: NC Expected With SMA | 0 | 3 | 0 | 1
  Week 13: NC Besides Those Expected With SMA | 0 | 0 | 0 | 0
  Week 13: NC Expected With SMA | 0 | 2 | 0 | 1
  Week 26: NC Besides Those Expected With SMA | 0 | 1 | 0 | 1
  Week 26: NC Expected With SMA | 10 | 52 | 45 | 4
  Week 39: NC Besides Those Expected With SMA | 0 | 0 | 0 | 1
  Week 39: NC Expected With SMA | 0 | 1 | 0 | 1
  Week 52: NC Besides Those Expected With SMA | 0 | 1 | 0 | 2
  Week 52: NC Expected With SMA | 11 | 65 | 61 | 10
  Week 61: NC Besides Those Expected With SMA | 0 | 0 | 0 | 0
  Week 61: NC Expected With SMA | 0 | 1 | 0 | 0
  Week 65: NC Besides Those Expected With SMA | 0 | 0 | 0 | 0
  Week 65: NC Expected With SMA | 0 | 2 | 0 | 1
  Week 78: NC Besides Those Expected With SMA | 0 | 1 | 0 | 2
  Week 78: NC Expected With SMA | 11 | 58 | 63 | 12
  Week 87: NC Besides Those Expected With SMA | 0 | 0 | 0 | 0
  Week 87: NC Expected With SMA | 0 | 1 | 0 | 0
  Week 91: NC Besides Those Expected With SMA | 0 | 0 | 0 | 1
  Week 91: NC Expected With SMA | 0 | 2 | 0 | 0
  Week 104: NC Besides Those Expected With SMA | 0 | 1 | 0 | 1
  Week 104: NC Expected With SMA | 11 | 64 | 63 | 12
  Week 130: NC Besides Those Expected With SMA | 0 | 0 | 0 | 1
  Week 130: NC Expected With SMA | 10 | 63 | 60 | 12
  Week 156: NC Besides Those Expected With SMA | 1 | 0 | 0 | 0
  Week 156: NC Expected With SMA | 7 | 62 | 57 | 12
  Week 169: NC Besides Those Expected With SMA | 0 | 0 | 0 | 0
  Week 169: NC Expected With SMA | 0 | 1 | 0 | 0
  Week 182: NC Besides Those Expected With SMA | 0 | 3 | 0 | 0
  Week 182: NC Expected With SMA | 9 | 52 | 55 | 9
  Week 208: NC Besides Those Expected With SMA | 0 | 2 | 1 | 0
  Week 208: NC Expected With SMA | 7 | 52 | 51 | 10
  Week 234: NC Besides Those Expected With SMA | 0 | 0 | 0 | 0
  Week 234: NC Expected With SMA | 10 | 53 | 50 | 9
  Week 260: NC Besides Those Expected With SMA | 0 | 0 | 0 | 0
  Week 260: NC Expected With SMA | 10 | 52 | 49 | 7

5. Primary Outcome: Number of Participants With Emergence or Worsening of Symptoms as Assessed Using Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS was used to assess the lifetime suicidality of a participant (baseline) as well as any new instances of suicidality (since last visit). The interview prompts recollection of suicidal ideation (SI), including the intensity of the ideation, behavior and attempts with actual/potential lethality. A modified and reduced version (pediatric version) was used for children (aged 6-11 years). Categories have binary responses (yes/no) & include: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active SI with Any Methods (Not Plan) without Intent to Act; Active SI with Some Intent to Act, without Specific Plan; Active SI with Specific Plan & Intent, Preparatory Acts & Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. SI or behavior is indicated by a "yes" answer to any of the listed categories. A score of 0 is assigned if no suicide risk is present. A score of 1 or higher indicates SI or behavior.
Time Frame: Up to approximately 5 years
Population: SE population included all participants who received at least one dose of risdiplam, whether prematurely withdrawn from the study or not. Participants with SI, suicidal behavior, and self-injurious behavior without suicidal intent are reported for this outcome measure. Overall number analyzed are the number of participants with at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101
Number analyzed (Participants) | 12 | 68 | 68 | 10
Participants
  Suicidal Ideation | 1 | 5 | 2 | 0
  Suicidal Behaviour | 0 | 0 | 0 | 0
  Self-injurious Behavior Without Suicidal Intent | 0 | 0 | 1 | 0

6. Primary Outcome: Anthropometric Examination: Change From Baseline in Weight
Description: Weight was measured at baseline, Weeks 65, 91, and every 13 weeks thereafter for participants 2-17 years and at every visit for participants <2 years. Per protocol, height was not measured at Day 7, Weeks 8, 17, 35, and thus not collected for all participants. No participants in the RO6885247 arm attended the Weeks 65, 169, 195, and 247 visit; none in the AVXS-101 arm attended the Week 247 visit. Symptom-directed height/weight assessments were done at clinically indicated visits as needed.
Time Frame: Baseline up to Week 260
Population: SE population included all participants who received at least one dose of risdiplam, whether prematurely withdrawn from the study or not. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101
Number analyzed (Participants) | 13 | 76 | 70 | 14
kilograms (kg)
  Baseline | 59.19 (20.47) | 39.29 (22.30) | 46.48 (15.57) | 12.87 (3.35)
  Day 7: number analyzed (Participants) | 9 | 3 | 0 | 0
  Day 7 | 0.09 (0.20) | 0.13 (0.31) |  |
  Week 2: number analyzed (Participants) | 13 | 75 | 69 | 13
  Week 2 | -2.79 (10.66) | 0.15 (0.80) | 0.19 (1.73) | 0.00 (0.32)
  Week 4: number analyzed (Participants) | 13 | 73 | 68 | 14
  Week 4 | -0.89 (3.15) | 0.29 (0.91) | 0.37 (1.86) | 0.03 (0.37)
  Week 8: number analyzed (Participants) | 9 | 3 | 0 | 0
  Week 8 | -0.17 (2.38) | 0.00 (0.17) |  |
  Week 13: number analyzed (Participants) | 2 | 63 | 62 | 9
  Week 13 | 0.45 (1.91) | 0.64 (1.57) | 0.63 (2.28) | 0.07 (0.46)
  Week 17: number analyzed (Participants) | 9 | 3 | 0 | 0
  Week 17 | -0.33 (2.91) | 2.07 (3.09) |  |
  Week 26: number analyzed (Participants) | 10 | 50 | 40 | 7
  Week 26 | -1.26 (3.99) | 1.25 (2.01) | 1.14 (4.03) | 0.52 (0.68)
  Week 35: number analyzed (Participants) | 9 | 6 | 4 | 0
  Week 35 | -1.51 (4.21) | 2.12 (1.69) | -0.10 (3.36) |
  Week 39: number analyzed (Participants) | 2 | 44 | 28 | 10
  Week 39 | -0.20 (2.55) | 1.06 (2.96) | 0.99 (2.68) | 0.90 (1.02)
  Week 43: number analyzed (Participants) | 9 | 8 | 7 | 2
  Week 43 | -1.09 (4.17) | 2.95 (3.92) | 1.56 (5.29) | 4.75 (3.32)
  Week 52: number analyzed (Participants) | 10 | 57 | 53 | 13
  Week 52 | -0.26 (3.32) | 1.93 (3.84) | 1.35 (3.39) | 1.71 (2.13)
  Week 61: number analyzed (Participants) | 1 | 7 | 6 | 1
  Week 61 | 6.40 (NA) — The standard deviation (SD) was not estimable for 1 participant. | 2.07 (1.70) | 0.25 (1.46) | 1.30 (NA) — The SD was not estimable for 1 participant.
  Week 65: number analyzed (Participants) | 0 | 43 | 46 | 10
  Week 65 |  | 2.96 (3.14) | 1.96 (3.87) | 2.54 (2.40)
  Week 70: number analyzed (Participants) | 6 | 4 | 3 | 1
  Week 70 | -1.72 (4.27) | -0.93 (3.97) | -1.38 (3.60) | 1.30 (NA) — The SD was not estimable for 1 participant.
  Week 78: number analyzed (Participants) | 9 | 57 | 59 | 14
  Week 78 | -0.19 (3.81) | 3.42 (3.84) | 1.77 (4.31) | 2.61 (2.37)
  Week 87: number analyzed (Participants) | 1 | 2 | 8 | 2
  Week 87 | 2.15 (NA) — The SD was not estimable for 1 participant. | 2.80 (4.67) | 3.91 (4.37) | 5.30 (5.80)
  Week 91: number analyzed (Participants) | 2 | 52 | 44 | 10
  Week 91 | -0.85 (3.68) | 4.33 (4.75) | 2.11 (4.99) | 2.07 (0.92)
  Week 96: number analyzed (Participants) | 1 | 5 | 16 | 1
  Week 96 | 9.60 (NA) — The SD was not estimable for 1 participant. | 3.52 (3.12) | 3.19 (4.98) | 0.70 (NA) — The SD was not estimable for 1 participant.
  Week 104: number analyzed (Participants) | 10 | 63 | 55 | 13
  Week 104 | 0.45 (4.50) | 3.96 (5.33) | 3.21 (5.02) | 3.08 (3.18)
  Week 117: number analyzed (Participants) | 1 | 12 | 10 | 5
  Week 117 | -0.10 (NA) — The SD was not estimable for 1 participant. | 4.30 (3.10) | 3.45 (3.24) | 1.86 (0.84)
  Week 130: number analyzed (Participants) | 9 | 58 | 56 | 13
  Week 130 | -0.60 (3.56) | 5.30 (6.07) | 2.95 (5.51) | 3.19 (1.49)
  Week 143: number analyzed (Participants) | 1 | 8 | 4 | 1
  Week 143 | 2.90 (NA) — The SD was not estimable for 1 participant. | 2.69 (4.04) | 4.35 (4.90) | 1.70 (NA) — The SD was not estimable for 1 participant.
  Week 156: number analyzed (Participants) | 10 | 59 | 56 | 12
  Week 156 | 0.28 (4.66) | 6.44 (6.39) | 3.81 (6.45) | 4.02 (2.10)
  Week 169: number analyzed (Participants) | 0 | 6 | 2 | 1
  Week 169 |  | 3.29 (5.49) | 8.90 (4.38) | 2.10 (NA) — The SD was not estimable for 1 participant.
  Week 182: number analyzed (Participants) | 9 | 53 | 56 | 10
  Week 182 | 1.94 (4.09) | 7.37 (6.96) | 4.27 (7.81) | 4.97 (2.41)
  Week 195: number analyzed (Participants) | 0 | 1 | 1 | 2
  Week 195 |  | 22.00 (NA) — The SD was not estimable for 1 participant. | 7.50 (NA) — The SD was not estimable for 1 participant. | 5.20 (0.99)
  Week 208: number analyzed (Participants) | 7 | 54 | 52 | 10
  Week 208 | 0.51 (2.68) | 8.70 (7.71) | 4.82 (8.37) | 5.44 (3.33)
  Week 221: number analyzed (Participants) | 2 | 1 | 1 | 1
  Week 221 | 1.35 (0.49) | 7.70 (NA) — The SD was not estimable for 1 participant. | 3.50 (NA) — The SD was not estimable for 1 participant. | 3.80 (NA) — The SD was not estimable for 1 participant.
  Week 234: number analyzed (Participants) | 9 | 51 | 48 | 8
  Week 234 | 1.56 (2.65) | 9.26 (7.91) | 6.29 (8.55) | 7.77 (5.04)
  Week 247: number analyzed (Participants) | 0 | 4 | 1 | 0
  Week 247 |  | 4.73 (4.89) | 11.10 (NA) — The SD was not estimable for 1 participant. |
  Week 260: number analyzed (Participants) | 10 | 52 | 48 | 7
  Week 260 | 2.81 (3.49) | 10.03 (8.41) | 7.41 (9.11) | 9.54 (6.23)

7. Primary Outcome: Anthropometric Examination: Change From Baseline in Height
Description: Height of all participants able to stand was measured while standing using a stadiometer, with at least 3 independent measurements, which were averaged. Participants unable to stand during the measurement, height was derived from measurement of ulna length. For very young children, height was measured with child in a lying position using an inflexible length board with fixed headboard & movable footboard. Height was measured: baseline, Weeks 13,39,52,78 & 104 for participants 2-17 years; Weeks 52 & 104 for >17 years & every visit for participants <2 years. After Week 104, measurements occurred every 26 weeks. Per protocol, height was not measured at Weeks 2,4,17,26,35,43,61,65,87,91,96,117,143,169,195,221 &247 & thus not collected for all participants. No participants <17 years in RO6885247, Olesoxime, or AVXS-101 arms attended the Week 260 visit & no participants in RO6885247 arm attended Week 39. Symptom-directed height assessments were done at clinically indicated visits as needed.
Time Frame: Baseline up to Week 260
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101
Number analyzed (Participants) | 13 | 76 | 70 | 14
centimeters (cm)
  Baseline: number analyzed (Participants) | 13 | 76 | 69 | 14
  Baseline | 171.36 (8.36) | 141.21 (26.17) | 161.71 (13.86) | 92.37 (11.23)
  Week 2: number analyzed (Participants) | 0 | 3 | 0 | 2
  Week 2 |  | 0.00 (0.00) |  | 0.00 (0.00)
  Week 4: number analyzed (Participants) | 0 | 2 | 0 | 3
  Week 4 |  | 1.00 (1.41) |  | 0.33 (0.58)
  Week 13: number analyzed (Participants) | 3 | 47 | 50 | 9
  Week 13 | -0.20 (1.71) | 1.08 (4.10) | 1.23 (5.09) | 2.78 (2.14)
  Week 17: number analyzed (Participants) | 6 | 3 | 0 | 0
  Week 17 | -0.84 (3.56) | -10.99 (28.36) |  |
  Week 26: number analyzed (Participants) | 0 | 2 | 0 | 2
  Week 26 |  | 6.50 (6.36) |  | 0.00 (1.41)
  Week 35: number analyzed (Participants) | 6 | 4 | 3 | 0
  Week 35 | -0.40 (3.75) | 2.92 (3.38) | 0.05 (1.25) |
  Week 39: number analyzed (Participants) | 0 | 30 | 13 | 8
  Week 39 |  | 4.81 (4.13) | 6.18 (9.33) | 2.41 (3.25)
  Week 43: number analyzed (Participants) | 0 | 5 | 2 | 1
  Week 43 |  | 11.41 (7.59) | 3.55 (5.01) | 7.00 (NA) — The SD was not estimable for 1 participant.
  Week 52: number analyzed (Participants) | 9 | 49 | 41 | 8
  Week 52 | -0.38 (2.98) | 6.14 (5.31) | 2.36 (5.66) | 6.83 (3.01)
  Week 61: number analyzed (Participants) | 1 | 3 | 3 | 0
  Week 61 | 0.00 (NA) — The SD was not estimable for 1 participant. | 11.41 (9.06) | 4.61 (6.33) |
  Week 65: number analyzed (Participants) | 0 | 7 | 3 | 3
  Week 65 |  | 9.80 (6.91) | 0.88 (0.76) | 8.00 (1.73)
  Week 78: number analyzed (Participants) | 3 | 50 | 49 | 10
  Week 78 | -0.71 (2.16) | 9.92 (6.32) | 3.90 (6.80) | 9.09 (4.04)
  Week 87: number analyzed (Participants) | 0 | 0 | 3 | 1
  Week 87 |  |  | 4.77 (3.05) | 5.78 (NA) — The SD was not estimable for 1 participant.
  Week 91: number analyzed (Participants) | 0 | 2 | 0 | 2
  Week 91 |  | 17.00 (7.07) |  | 10.00 (4.24)
  Week 96: number analyzed (Participants) | 0 | 0 | 7 | 0
  Week 96 |  |  | 6.96 (14.28) |
  Week 104: number analyzed (Participants) | 8 | 57 | 47 | 11
  Week 104 | -0.87 (1.92) | 11.33 (7.14) | 5.14 (7.33) | 14.54 (3.95)
  Week 117: number analyzed (Participants) | 0 | 4 | 2 | 0
  Week 117 |  | 9.20 (6.11) | 4.86 (3.15) |
  Week 130: number analyzed (Participants) | 5 | 50 | 48 | 10
  Week 130 | -1.60 (2.13) | 12.15 (8.73) | 4.70 (7.80) | 16.11 (5.48)
  Week 143: number analyzed (Participants) | 1 | 3 | 1 | 0
  Week 143 | 0.00 (NA) — The SD was not estimable for 1 participant. | 5.91 (6.39) | 5.00 (NA) — The SD was not estimable for 1 participant. |
  Week 156: number analyzed (Participants) | 5 | 47 | 46 | 9
  Week 156 | -0.20 (0.45) | 12.90 (10.31) | 4.43 (6.80) | 22.02 (4.97)
  Week 169: number analyzed (Participants) | 0 | 3 | 1 | 0
  Week 169 |  | 13.46 (12.09) | 0.00 (NA) — The SD was not estimable for 1 participant. |
  Week 182: number analyzed (Participants) | 6 | 41 | 43 | 7
  Week 182 | -2.25 (5.54) | 15.36 (11.34) | 4.67 (6.31) | 21.54 (2.76)
  Week 195: number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 195 |  |  |  | 31.74 (NA) — The SD was not estimable for 1 participant.
  Week 208: number analyzed (Participants) | 6 | 44 | 36 | 7
  Week 208 | -2.28 (5.52) | 16.13 (11.69) | 4.91 (8.60) | 26.17 (6.55)
  Week 221: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 221 | 0.00 (NA) — The SD was not estimable for 1 participant. |  | 9.77 (NA) — The SD was not estimable for 1 participant. |
  Week 234: number analyzed (Participants) | 8 | 41 | 34 | 6
  Week 234 | -1.04 (5.25) | 17.18 (13.14) | 4.95 (7.88) | 28.21 (5.49)
  Week 247: number analyzed (Participants) | 0 | 2 | 0 | 0
  Week 247 |  | 10.18 (14.39) |  |
  Week 260: number analyzed (Participants) | 0 | 2 | 0 | 0
  Week 260 |  | 29.00 (5.66) |  |

8. Primary Outcome: Anthropometric Examination: Change From Baseline in Head Circumference
Description: Head circumference for participants aged < 5 years was measured to the nearest 0.1 cm using a flexible, non-stretchable tape. Head circumference was measured around the widest part of the head from the most prominent point on the back of the head (occiput) to the most prominent part of the forehead between the eyebrows. The measurement was repeated three times, and the largest measurement was recorded. Head circumference was assessed for participants < 5 years of age. Since all participants in the RO6885247 and Olesoxime arms were > 5 years, data were not collected for these arms. Head circumference was not collected at Weeks 35 and 61 (AVXS-101 arm) and Weeks 87, 182, and 208 (Nusinersen arm) because the protocol only required this measurement for participants < 5 years of age. At these timepoints, neither of the participants < 5 years attended the visit, and other participants may have been > 5 years of age.
Time Frame: Baseline up to Week 208
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101
Number analyzed (Participants) | 0 | 10 | 0 | 14
cm
  Baseline: number analyzed (Participants) | 0 | 10 | 0 | 13
  Baseline |  | 51.10 (3.43) |  | 50.61 (2.15)
  Week 2: number analyzed (Participants) | 0 | 6 | 0 | 12
  Week 2 |  | 0.28 (0.85) |  | 0.26 (0.43)
  Week 4: number analyzed (Participants) | 0 | 6 | 0 | 13
  Week 4 |  | 0.27 (1.55) |  | 0.17 (0.51)
  Week 13: number analyzed (Participants) | 0 | 4 | 0 | 8
  Week 13 |  | 0.70 (1.54) |  | 0.51 (0.51)
  Week 26: number analyzed (Participants) | 0 | 4 | 0 | 5
  Week 26 |  | 1.30 (0.77) |  | 0.58 (1.02)
  Week 35: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 35 |  | 0.00 (NA) — The SD was not estimable for 1 participant. |  |
  Week 39: number analyzed (Participants) | 0 | 3 | 0 | 6
  Week 39 |  | 1.90 (1.15) |  | 0.42 (0.99)
  Week 52: number analyzed (Participants) | 0 | 3 | 0 | 8
  Week 52 |  | 1.90 (1.15) |  | 1.34 (0.91)
  Week 61: number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 61 |  | 1.50 (NA) — The SD was not estimable for 1 participant. |  |
  Week 65: number analyzed (Participants) | 0 | 2 | 0 | 3
  Week 65 |  | 2.75 (1.77) |  | 1.67 (1.89)
  Week 78: number analyzed (Participants) | 0 | 3 | 0 | 8
  Week 78 |  | 2.40 (1.44) |  | 1.58 (0.75)
  Week 87: number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 87 |  |  |  | 0.50 (NA) — The SD was not estimable for 1 participant.
  Week 91: number analyzed (Participants) | 0 | 1 | 0 | 2
  Week 91 |  | 1.50 (NA) — The SD was not estimable for 1 participant. |  | 1.05 (2.05)
  Week 104: number analyzed (Participants) | 0 | 2 | 0 | 7
  Week 104 |  | 1.60 (0.14) |  | 1.70 (0.77)
  Week 130: number analyzed (Participants) | 0 | 1 | 0 | 6
  Week 130 |  | 5.50 (NA) — The SD was not estimable for 1 participant. |  | 2.10 (1.52)
  Week 156: number analyzed (Participants) | 0 | 1 | 0 | 2
  Week 156 |  | 3.00 (NA) — The SD was not estimable for 1 participant. |  | 3.00 (0.71)
  Week 182: number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 182 |  |  |  | 3.50 (NA) — The SD was not estimable for 1 participant.
  Week 208: number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 208 |  |  |  | 3.50 (NA) — The SD was not estimable for 1 participant.

9. Primary Outcome: Maximum Plasma Concentration (Cmax) of Risdiplam
Description: As pre-specified in the protocol, the PK data were not to be compared between participants who received different prior treatments (RO6885247, nusinersen, olesoxime and AVXS-101) received before entering this study, but to analyze the PK parameters of risdiplam. Hence, PK data have been presented in a single arm group irrespective of prior therapies received by the participants in previous studies.
Time Frame: Predose on Weeks 2, 4, 13, 26, 39, 52, 65, 91 and post-dose on Weeks 1, 4, 13, 52, 91 and 104
Population: PK population included all participants with at least one timepoint with a measurable drug concentration. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: nanograms per milliliter (ng/mL)
Groups:
- Risdiplam: Participants previously treated with the splicing modifier, RO6885247 or placebo in study BP29420, or participants treated with nusinersen, olesoxime and AVXS-101 received risdiplam, PO, QD, based on their body weight and age during the 24-month treatment phase. After the 24-month treatment phase, participants who chose to enter the OLE phase continued receiving risdiplam, PO, QD, based on their body weight and age up to a maximum of 3 years.
Arm/Group | Risdiplam
Number analyzed (Participants) | 173
nanograms per milliliter (ng/mL) | 120 [38.1 to 258]

10. Primary Outcome: Area Under the Concentration-Time Curve (AUC0-24h) of Risdiplam
Description: as for outcome 9
Time Frame: 24 hours Postdose at Year 2 Visit
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Risdiplam
Number analyzed (Participants) | 122
nanograms*hour/milliliter (ng*h/mL) | 1720 [983 to 2670]

11. Primary Outcome: Plasma Trough Concentration (Ctrough) of Risdiplam
Description: as for outcome 9
Time Frame: Predose at Year 5 visit
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Risdiplam
Number analyzed (Participants) | 113
ng/mL | 57.5 [17.7 to 168]

12. Secondary Outcome: Survival of Motor Neuron (SMN) Protein Levels in Blood
Description: SMA is caused by a homozygous deletion or mutation of the SMN 1 gene, which encodes SMN, an essential protein expressed in both neuronal and non-neuronal cells. In humans, there are two SMN genes, the SMN1 gene and its paralog SMN2. Risdiplam directly targets the underlying molecular deficiency of the disease and promotes the inclusion of exon 7 to generate full-length SMN2 mRNA, which therefore increases the production of functional SMN protein. As pre-specified in the protocol, the PD data were not to be compared between participants who received different prior treatments, but to analyze the PD parameters of risdiplam. Hence, PD data have been presented in a single arm group irrespective of prior therapies received by the participants in previous studies.
Time Frame: Baseline and Year 5
Population: Pharmacodynamic (PD) population included all participants with at least one timepoint with a measurable PD marker. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Risdiplam
Number analyzed (Participants) | 147
ng/mL
  Baseline | 3.35 [0.527 to 8.16]
  Year 5 | 6.51 [0.497 to 13.4]

ADVERSE EVENTS:
Time Frame: Up to approximately 5 years
Description: SE population included all participants who received at least one dose of risdiplam, whether prematurely withdrawn from the study or not. 1 participant previously treated with 'Olesoxime' discontinued per physician's decision before receiving any treatment and was not included in SE population. As pre-planned, data for the treatment and OLE phases were collected and reported together, since participants received the same dose of risdiplam throughout the study.
Arm/Group | RO6885247 | Nusinersen | Olesoxime | AVXS-101
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/76 | 0/70 | 2/14
Serious Adverse Events (participants affected / at risk) | 3/13 | 25/76 | 24/70 | 8/14
Other Adverse Events (participants affected / at risk) | 12/13 | 76/76 | 69/70 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO6885247 (N=13) | Nusinersen (N=76) | Olesoxime (N=70) | AVXS-101 (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal muscular atrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blindness transient (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (4) | 2 (3) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Metapneumovirus pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 4 (7) | 5 (6) | 1 (2)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Incision site impaired healing (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO6885247 (N=13) | Nusinersen (N=76) | Olesoxime (N=70) | AVXS-101 (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 8 (10) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 5 (7) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 6 (6) | 5 (11) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (5) | 7 (11) | 2 (3)
Aphthous ulcer (Gastrointestinal disorders) | 2 (3) | 7 (11) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (7) | 4 (7) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 20 (23) | 12 (22) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (6) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 14 (24) | 9 (16) | 1 (1)
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 10 (15) | 12 (21) | 7 (23)
Cyst (General disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 11 (13) | 5 (5) | 0 (0)
Feeling jittery (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 2 (2) | 4 (5) | 2 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 3 (7) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 28 (51) | 14 (20) | 9 (22)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dust allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 8 (13) | 11 (20) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 28 (31) | 28 (34) | 3 (4)
Cellulitis (Infections and infestations) | 0 (0) | 4 (7) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 1 (2) | 4 (5) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 4 (5) | 3 (3) | 3 (3)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 14 (15) | 5 (7) | 3 (4)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 9 (11) | 6 (10) | 2 (3)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (3) | 2 (2) | 0 (0)
Metapneumovirus pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 17 (38) | 16 (28) | 8 (18)
Otitis media (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 5 (5) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1) | 6 (9) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 7 (11) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 4 (6) | 3 (3) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 21 (45) | 22 (34) | 7 (16)
Urinary tract infection (Infections and infestations) | 2 (16) | 6 (9) | 7 (7) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 9 (13) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 4 (5) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 7 (8) | 3 (6) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 3 (4)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Human metapneumovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (3) | 1 (1) | 4 (4) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary sediment present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (10) | 9 (14) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 6 (6) | 6 (13) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 6 (10) | 4 (5) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 21 (42) | 17 (51) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (6) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 6 (6) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Procedural anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (4) | 3 (5) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (3) | 4 (5) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (8) | 0 (0)
Strangury (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 9 (23) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 17 (25) | 10 (12) | 4 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (3) | 2 (3)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (8) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 7 (10) | 11 (16) | 2 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (4) | 1 (1)
Sleep-related hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 5 (7) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 5 (7) | 0 (0)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 11 (11) | 7 (8) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria aquagenic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyanosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03032172/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT03032172/SAP_001.pdf